CLINICAL TRIAL: NCT05868369
Title: The Effectiveness of Immersive Virtual Reality as a Pain Control Modality After Hip Arthroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michael Banffy, MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002535
Record Dates: First submitted 2023-02-28; First posted 2023-05-22 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hip Pain Chronic
Keywords: virtual reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard regimen +iVR Group (Experimental): postoperative iVR therapy in addition to the standard multimodal pain regimen (including a preoperative local field block
  Interventions: Device: iVR Group; Drug: Standard pain management regimen
- Standard regimen (Active Comparator): hip arthroscopy patients who receive only the standard regimen (including field block) in the acute postoperative ambulatory setting
  Interventions: Drug: Standard pain management regimen

INTERVENTIONS:
Device: iVR Group — On the day of surgery, the iVR group will receive a 30-minute sessions or "dose" of iVR therapy in the ambulatory post-anesthesia care unit (PACU) during their stay. The three distraction-based or skills-based iVR modules will consist of either 1) Mindful Escape; 2) Empowered Breathing; or 3) Relaxation videos. The iVR group will be sub-randomized into receiving only one of the three types of modules. The modules will start approximately 30 minutes upon arriving in PACU and will last approximately 30 minutes.
  Arms: Standard regimen +iVR Group
Drug: Standard pain management regimen — In the ambulatory post-anesthesia care unit (PACU) during their stay with have standard postoperative pain protocol (including a pre-operative local field block).

SUMMARY:
1. The purpose of the research is to assess the efficacy of postoperative immersive virtual reality (iVR) compared to a standard multimodal pain regimen including opioids and a local block on acute postoperative pain management following hip arthroscopy
2. The primary research procedures are medical record review for demographic information, head-mounted immersive virtual reality experience in PACU, and pre-operative and post-operative surveys
3. The study will enroll adult patients of all ages undergoing elective hip arthroscopy procedures for any diagnosis

DETAILED DESCRIPTION:
The overall purpose of this prospective matched cohort investigation is to assess the efficacy of postoperative iVR compared to a standard multimodal pain regimen including opioids, on acute postoperative pain management following hip arthroscopy. The goal is to determine whether iVR in the immediate post-operative ambulatory setting would have any effect on subjective pain, anxiety, and nausea scores or on patients' opioid consumption. The primary objective of this study is to evaluate the effects of administering a head-mounted immersive virtual reality (iVR) experience to control postoperative pain and nausea in patients undergoing hip arthroscopy. The secondary objective of this study is to evaluate the effectiveness of specific iVR modules in pain perception and decreasing overall opioid use for post-operative pain control. We will prospectively compare a cohort of primary hip arthroscopy patients who receive postoperative iVR therapy in addition to the standard multimodal pain regimen (including a preoperative local field block) with a matched cohort of hip arthroscopy patients who receive only the standard regimen (including field block) in the acute postoperative ambulatory setting. On the day of surgery, the iVR group will receive a 30-minute sessions or "dose" of iVR therapy in the ambulatory post-anesthesia care unit (PACU) during their stay in addition to the standard postoperative pain protocol (including a pre-operative local field block). The three distraction-based or skills-based iVR modules will consist of either 1) Mindful Escape; 2) Empowered Breathing; or 3) Relaxation videos. The iVR group will be sub-randomized into receiving only one of the three types of modules. The modules will start approximately 30 minutes upon arriving in PACU and will last approximately 30 minutes. Both groups will receive the standard postoperative pain protocol on an as needed basis.

The duration of the study is three weeks (pre-operative visit, operative day, and first post-operative visit).

Patients will be screened and enrolled at their pre-operative visit. Included patients will be consented and will fill out the pre-operative questionnaires in order to provide baseline data. They will be randomized into the control group or the iVR therapy group. On the day of surgery, they will undergo their local field block by their anesthesiologist pre-operatively, undergo their hip arthroscopy procedure as indicated by their surgeon, and undergo their VR therapy in PACU as described above. They will be asked for their pain scores when leaving PACU, and their opioid medication usage during PACU will be recorded. Post-operative questionnaires will also be completed prior to discharge from PACU and at the first post-op visit.

The study involves participation at a single timepoint only. The study procedures to be done are listed below: Virtual Reality Therapy in PACU performed once as described above.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with hip pathology
* Failed non-operative treatment of hip pathology
* Undergoing primary, elective and isolated hip arthroscopy for their hip pathology
* Complete pre-operative and post-operative questionnaires

Exclusion Criteria:

* Minors (17 years of age and younger)
* Traumatic injuries undergoing emergent surgery
* Undergoing revision hip arthroscopic surgery
* Do not complete pre-operative and post-operative questionnaires
* Patients not able to undergo elective surgery
* Pregnant women
* Prisoners
* Patients with conditions that interfere with VR usage including: history of seizure or epilepsy, facial injury precluding safe placement of headset, visual impairment impacting ability to visualize VR images, hearing impairment impacting ability to follow audio instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Pain visual analog scale (VAS) | one time at Day 1 post operative
  subjects rate their pain from 0-10, 0 being the least and 10 being the worst.

SECONDARY OUTCOMES:
Anxiety PACU questionnaire | one time Day 1 of surgery post-op
  On a scale 1-9 1 being the least and 9 being the worst
Nausea PACU Questionnaire | one time Day 1 of surgery post-op
  On a scale none, slight, moderate and sever.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ladnier, MS, Study Director — Cedar -Sinai Kerlan jobe orthopedic institute
Locations (1):
- Kerlan Jobe, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No